CLINICAL TRIAL: NCT06973434
Title: "Effects of Conventional and Video Laryngoscopy Methods on VIDIAC Scores and Hemodynamic Stability in Obese Patients: Comparison of Storz C-MAC3, Scoper MAC-3 and Macintosh"
Brief Title: Comparison of Video and Direct Laryngoscopy in Obese Patients During Surgery
Status: Recruiting | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veli Fahri Pehlivan, Assistant Professor, Harran University
Other Study IDs: Ümit
Record Dates: First submitted 2025-04-10; First posted 2025-05-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Obesity Difficult Airway Airway Management
Keywords: Video laryngoscopy; Obesity; VIDIAC score; Storz C-MAC; Scoper MAC
MeSH Terms: conditions — Obesity | interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 (n=40) Intubated with Storz C-MAC3 video laryngoscope: Participants in this group will be intubated using the Storz C-MAC3 video laryngoscope. Preoperative difficult intubation risk, and pre- and post-induction vital signs (heart rate, systolic and diastolic blood pressure, mean arterial pressure) will be recorded. Additionally, VIDIAC scores specific to video-assisted intubation and early postoperative intubation complications will be assessed for this group.
  Interventions: Device: intubation
- Group 2 (n=40): Intubated with Scoper MAC-3 video laryngoscope: Participants in this group will be intubated using the Scoper MAC-3 video laryngoscope. Preoperative difficult intubation assessment, pre- and post-induction hemodynamic parameters (heart rate, systolic and diastolic blood pressure, mean arterial pressure), VIDIAC scoring for video laryngoscopy, and postoperative airway-related complications will be evaluated.
  Interventions: Device: intubation
- Group 3 (n=40): Control group intubated with Macintosh laryngoscope: Participants in the control group will be intubated using a standard Macintosh direct laryngoscope. Their preoperative airway risk, vital signs before and after induction, and intubation-related complications will be recorded. VIDIAC score will not be used for this group as it applies only to video laryngoscopy.
  Interventions: Device: intubation

INTERVENTIONS:
Device: intubation — intubation

SUMMARY:
This study aims to evaluate how intubation performed with two different brands of videolaryngoscope and the Macintosh laryngoscope during surgeries in obese patients requiring general anesthesia affects the VIDIAC score, hemodynamic response, and early postoperative complications. Complications such as sore throat, hoarseness, nausea, and vomiting will be recorded in the recovery room prior to discharge.

DETAILED DESCRIPTION:
Success in airway management is critical for the safety of anesthesia practices. Unsuccessful airway management is a leading cause of anesthesia-related morbidity-including airway trauma, dental injury, pulmonary aspiration, unplanned tracheostomy, hypoxic brain injury, and cardiopulmonary arrest-and mortality.

Unsuccessful airway management accounts for approximately 30-40% of anesthesia-related deaths. In a review of closed insurance claims against anesthesiologists, 17% were related to difficult or impossible intubation without documented preoperative airway assessment.

Video laryngoscopes are technological tools used to visualize airway structures and facilitate endotracheal intubation, particularly in patients with anticipated difficult airways.

Obesity is a metabolic disorder characterized by excessive fat accumulation and is associated with both physical and psychological complications. It is an independent risk factor for difficult airway and increases the risk of anesthesia-related complications. Obesity is also linked to restrictive lung disease due to increased intra-abdominal pressure and decreased thoracic compliance. The resulting reductions in static and dynamic lung volumes lead to rapid desaturation during apnea or hypoventilation, primarily due to reduced functional residual capacity and expiratory reserve volume.

In this prospective observational study, the investigators aim to perform a comparative analysis of VIDIAC scores, hemodynamic responses (heart rate, systolic and diastolic blood pressure, mean arterial pressure), and early postoperative complications following laryngoscopy performed with Storz C-MAC videolaryngoscope, Scoper videolaryngoscope, and Macintosh laryngoscope in obese patients undergoing elective surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Body mass index (BMI) ≥30 kg/m²
* ASA physical status I or II
* Scheduled for elective surgery
* Requiring endotracheal intubation
* Provided written informed consent

Exclusion Criteria:

* Refusal to participate in the study
* ASA physical status III, IV, or V
* Advanced cardiopulmonary disease
* Cervical spine movement limitation
* Pregnancy
* Coagulopathy
* Emergency surgery indication
* Known or anticipated difficult airway
* Severe anatomical deformity of the airway

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients between the ages of 18 and 65 years with a body mass index (BMI) of ≥30 kg/m², classified as American Society of Anesthesiologists (ASA) physical status I or II. All participants will be scheduled for elective surgery requiring general anesthesia and endotracheal intubation. Eligible participants must meet the inclusion criteria for obesity and provide written informed consent. Patients will be excluded if they have a known or anticipated difficult airway, advanced cardiopulmonary disease, pregnancy, coagulopathy, cervical spine movement limitation, or if they are scheduled for emergency surgery.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
VIDIAC (Video Intubation Difficulty Assessment and Classification) Score | Immediately after intubation (within 1 minute)
  Airway visualization will be assessed using the Video Intubation Difficulty Assessment and Classification (VIDIAC) scoring system during intubation. The VIDIAC score ranges from 1 to 5. A lower score indicates better visualization and easier intubation, while a higher score reflects increased difficulty. Score (1-5 scale)
Heart Rate Change | Baseline to 5 minutes post-intubation
  Change in heart rate from baseline (pre-induction) to 5 minutes after intubation

SECONDARY OUTCOMES:
Successful First-Attempt Intubation Rate | Immediately after intubation (within 1 minute)
  Proportion of patients successfully intubated on the first attempt using the assigned laryngoscope device.laryngoscope.
Intubation Time | Immediately after intubation
  Time measured in seconds from insertion of the laryngoscope blade to confirmation of successful endotracheal tube placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Veli Fahri Pehlivan, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No